CLINICAL TRIAL: NCT06552026
Title: Intermittent Theta Burst Stimulation on Anhedonia of Treatment Resistant Depression and Brian Network Mechanism
Brief Title: Intermittent Theta Burst Stimulation on Anhedonia in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fengqiong Yu, Professor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y&F
Record Dates: First submitted 2024-07-22; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Depression; Electroencephalography; Transcranial Magnetic Stimulation
Keywords: anhedonia; intermittent theta burst stimulation
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Intervention Model Description: a parallel two-arm model ,Participants were randomized to two groups by coin toss, and delivered rTMS or iTBS over the lDLPFC-NAcc once daily for 15 consecutive days.
Who Masked: Participant, Investigator
Masking Description: In this clinical trial, a double-blind design will be implemented. Neither the participants nor the researchers conducting the trial will be aware of the specific objectives or the allocation of treatment conditions. This approach is intended to eliminate bias and ensure the integrity of the study's outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iTBS stimulation (Experimental): The iTBS stimulation lasted 3 min 9 s and delivered at triplet 50 Hz bursts, repeated at 5 Hz with 2s on, 8 s off, 600 pulses per session at 80% of the rest motor threshold(RMT) . Behavior and EEG dataset should be acquired before the first iTBS session and after the last iTBS session.
  Interventions: Device: repeated transcranial magnetic stimulation
- 10 Hz-rTMS stimulation (Active Comparator): The rTMS stimulation lasted 25 mins and delivered at 10 Hz with 1s duration,4s rest, a total of 3000 pulses at 100% of the rest motor threshold(RMT) . Behavior and EEG dataset should be acquired before the first rTMS session and after the last rTMS session.
  Interventions: Device: repeated transcranial magnetic stimulation

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation — repetitive transcranial magnetic stimulation by use of high-frequency (10 Hz) left-side DLPFC stimulation is currently widely used in the treatment of depression17.Intermittent theta burst stimulation (iTBS) is a newer form of rTMS that can be delivered with shorter duration of stimulation sessions and apparent efficacy at lower stimulation intensities18. Both 10 Hz and intermittent theta burst stimulation pulses have an excitatory effect on cortical excitability

SUMMARY:
Study comparing the efficacy of two TMS patterns (intermittent theta-burst stimulation, iTBS, and repetitive transcranial magnetic stimulation, rTMS) in treating anhedonia and their associated brain network mechanisms.

DETAILED DESCRIPTION:
Anhedonia is a core feature in major depressive disorders, severely affecting up to 70% patients and remaining untreated after traditional antidepressants therapies. In previous work, the investigators provided clinical evidence for the therapeutic efficacy of personalized rTMS in treating anhedonia. However, the key practical question is whether personalized, connectivity-guided iTBS performs comparably to the existing standard rTMS about the clinical efficacy.

This study was designed as a double-blind controlled trial to investigate the intervention effect of iTBS stimulation on anhedonia in depressed patients. 33 subjects were included, 17 participated in conventional 10 Hz-rTMS treatment and 16 in iTBS treatment. Using the subjects' MRI imaging data of the nucleus accumbens (NAcc) as a seed point, individualized left dorsolateral prefrontal cortex (lDLPFC) targets were calculated from brain imaging data. Patients received once-daily treatment for 15 days.

Clinical symptoms, behavioral and EEG assessments were performed before and after treatment. Clinical assessments included The Hamilton Anxiety Scale (HAMA), the Hamilton Depression Rating Scale (HAMD), the Beck Depression Inventory (BDI), the Temporal Experience of Pleasure Scale (TEPS), and Apathy Evaluation Scale (AES); behavioral and EEG data were collected by the Monetary paradigm. One month after the end of the intervention, follow-up BDI, TEPS, and AES symptom data were collected by electronic scales. This study focused on the analysis of scale, behavioral, and EEG data of subjects .

ELIGIBILITY:
Inclusion Criteria:

diagnosed by more than two clinical psychiatrists, using the DSM-5 diagnostic criteria for depression.

the Self-Report Apathy Evaluation Scale score was more than 37 and the The Temporal Experience of Pleasure Scale score was less than 76.

consistent medical therapeutic plan for ≥4 weeks or no history of antidepressant drugs before rTMS treatment.

aged between 16 and 50 years old.

Exclusion Criteria:

participants with unstable physical conditions, pregnancy or those that were breastfeeding.

metal implants on or inside the head. increased intracranial pressure from cerebral infarction or brain injury. a history of substance abuse or major psychiatric diseases other than depression and current use of psychoactive drug.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms severity | Baseline;15 days after treatment
  The Hamilton depression rating scale-17 items (HAMD-17) to clinically assess severity of depression. The curative effects of the treatment were classified according to the reduction in HAMD. Response was defined as ≥50% symptom reduction from pre-to post-treatment with a HAMD score; remission criteria were set at a post-treatment score ≤7 for HAMD.
Change from baseline in Motivation and Pleasure Scale | Baseline;15 days after treatment
  Change from baseline in Motivation and Pleasure Scale The severity of participants' anhedonia assessed by the Motivation and Pleasure Scale change from baseline after the treatment.

SECONDARY OUTCOMES:
The alteration from baseline in electrophysiological source imaging results in multimodalities | Baseline;15 days after treatment
  The activation of nucleus accumbens, dorsal lateral prefrontal cortex and the functional connection these brain area assessed by source-level resting-state EEG connectivity in multimodalities change from baseline after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, PHD, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China